CLINICAL TRIAL: NCT02873910
Title: Randomized, Double-Blind, Placebo-Controlled, Monocentric, Parallel-Group Study to Evaluate the Influence of IQPAS-119 on Post-Marathon Susceptibility to Infections and Influence on Other Complaints and Its Tolerability: A Pilot Study
Brief Title: Influence of IQPAS-119 on Post-Marathon Susceptibility to Infections and Others
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InQpharm Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INQ/009716
Record Dates: First submitted 2016-08-08; First posted 2016-08-22 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2018-01

CONDITIONS: Upper Respiratory Tract Symptoms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- IQP-AS-119 (Experimental): One tablet to be taken daily with any meal, with a glass of water. They should not be chewed, but swallowed whole.
  Interventions: Dietary Supplement: IQP-AS-119
- Placebo (Placebo Comparator): One tablet to be taken daily with any meal, with a glass of water. They should not be chewed, but swallowed whole.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: IQP-AS-119
  Arms: IQP-AS-119
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the benefit and tolerability of IQP-AS-119 for reduction of susceptibility to infections and other complaints after extreme physical stress (participation in a marathon).

ELIGIBILITY:
Inclusion Criteria:

1. Caucasian males and females, 18-65 years of age, residents of Berlin or Brandenburg
2. Body mass index (BMI) 18.5-26.0 kg/m2
3. Registered as runner for the 43rd BMW Berlin Marathon 2016
4. History of at least 2 successful finished marathons (personal record of 3-5.5h within the last 5 years)
5. History of post-exercise susceptibility to infections (e.g. upper respiratory tract symptoms) and/or other health conditions (infections, stress complaints) after strenuous exercise (eg. marathon, half-marathon, bicycle races, triathlons, heavy training loads) within the last 5 years (to be distinctly documented at screening)
6. Readiness to comply with all study procedures, in particular:

   * Consumption of the investigational product (IP) during the entire treatment period of the study
   * Maintaining the habitual diet, with the exception of consumption of maximal 2 garlic cloves per week
   * Adapt pre-marathon training / physical activity to generally accepted proven or individually successful training plan
   * Adapt post-marathon training / physical activity to generally accepted proven or individually successful recovery plan
   * Filling in diaries and questionnaires
7. Readiness to ensure generally proven or individually successful optimal food intake and rehydration before, during, and after the marathon.
8. Non-smoker / smoking cessation of last ≥12 months prior to screening
9. Regular sleeping pattern (no suspicion of sleep disorder) in the three months prior to screening
10. Stable concomitant, permitted medication (if any) for at least last 2 weeks prior to screening and during the study
11. Women of child-bearing potential only:

    1. negative pregnancy testing (Beta human chorionic gonadotropin (ß-HCG) in urine) at screening
    2. commitment to use reliable contraception methods during the entire study

Participation is based upon written informed consent form (ICF) by the participant following written and oral information by the investigator regarding nature, purpose, consequences and possible risks of the clinical study.

Exclusion Criteria:

1. Known sensitivity to any ingredients of the IP
2. Additional strenuous exercise/activity other than regular occupational load, completing training runs / exercises prior the marathon. Additional strenuous exercise/activity other than regular occupational load and recovery exercise loads after the marathon
3. History of severe cardiovascular disease or collapse during a running event (half marathon, marathon etc.) and/or training
4. Hypertension (systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg)
5. Any abnormality observed in screening exercise ECG pointing to an increased cardiovascular risk (alternatively: any abnormality in the results of an exercise ECG performed in the last 6 weeks prior to screening pointing to an increased cardiovascular risk)
6. Any chronic disease affecting the upper respiratory tract and the lungs, eg. asthma bronchial, chronic obstructive pulmonary disease, or ears-nose-throat (ENT) infection
7. Acute infection of ENT or upper respiratory tract (URT) within the last month prior to screening
8. Any nasal abnormalities:

   1. History of nasal reconstructive surgery
   2. Severe nasal septum deviation or other condition that could cause nasal obstruction
   3. Presence of nasal ulcers or nasal polyps
9. Active organ or systemic diseases including severe cardiovascular disease, diabetes mellitus, renal or liver disorder
10. Known congenital or acquired immunodeficiency disease (e.g. HIV infection)
11. Known bleeding disorders such as bleeding ulcers, or haemophilia
12. Vaccination against influenza within 3 months prior to screening; any vaccination planned during the study
13. Anticoagulants such as warfarin
14. Systemic analgesics (other than paracetamol up to 2000mg/day or ibuprofen up to max. 800 mg/day, or if medically indicated and prescribed by a physician), antibiotics (unless medically indicated and prescribed by a physician) or decongestant nose drops / spray (except for isotonic sea water, or if medically indicated and prescribed by a physician) during the study
15. Use of medications or supplements influencing immune function (e.g. antihistamines, systemic corticosteroids, immune-suppressants), and physical performance, as per investigator's judgement, during the study
16. Use of any doping substance as listed by the "World Anti-Doping Agency" at present or in the past, unless prescribed by a physician under a '"therapeutic use exemption", per investigator's judgement
17. Any use of food supplements containing vitamins, minerals, or trace elements, as per investigator's judgement, during the study
18. Alcohol abuse (men: ≥21 units/week, women: ≥14 units/ week; 1 unit equals approximately 250 mL of beer, 100 mL of wine or 35 mL of spirits)
19. Women of child-bearing potential: pregnant or breastfeeding
20. Participation in other studies within the last month prior to screening and during study
21. Any other clinically significant condition which in the investigator's opinion could interfere with the results of the study or the safety of the subject

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2016-07-10 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2016-10-31 (Actual)

PRIMARY OUTCOMES:
Change in Hooper's Index | 5 weeks
  Compared between verum and placebo groups at baseline and all timepoints thereafter.

SECONDARY OUTCOMES:
Perceived Stress Questionnaire (PSQ20) | 5 weeks
  Compared between verum and placebo groups at baseline and all timepoints thereafter.
URT symptoms recorded in daily dairy | 5 weeks
  Compared between verum and placebo groups at baseline and all timepoints thereafter.
Daily subject diary on URT symptoms and other health conditions (including Overall Treatment Effect (OTE) | 5 weeks
  Compared between verum and placebo groups at baseline and all timepoints thereafter.
Wisconsin upper respiratory symptom survey (WURSS-21) | 5 weeks
  Compared between verum and placebo groups at baseline and all timepoints thereafter.
Short Form-12 (SF-12) Health Survey | 5 weeks
  Compared between verum and placebo groups at baseline and all timepoints thereafter.
Global evaluation of benefit (4-point categorical scale) | 5 weeks
  Measured by the subjects/investigator at the final visit only
Blood pressure | 5 weeks
  Compared between verum and placebo groups at baseline and all timepoints thereafter.
Pulse rate | 5 weeks
  Compared between verum and placebo groups at baseline and all timepoints thereafter.
Body temperature | 5 weeks
  Compared between verum and placebo groups at baseline and all timepoints thereafter.
Adverse events (AEs) throughout study | 5 weeks
  Compared between verum and placebo groups at baseline and all timepoints thereafter.
Global evaluation of tolerability (4-point categorical scale) | 5 weeks
  Measured by the subjects/investigator

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Uebelhack, MD, PhD, Principal Investigator — analyze & realize GmbH
Locations (1):
- analyze & realize GmbH, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No